CLINICAL TRIAL: NCT00000692
Title: Phase I Rising Dose Tolerability Study of SC-48334 in Patients With Acquired Immunodeficiency Syndrome (AIDS) and Advanced AIDS Related Complex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: G D Searle (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 100
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-03

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Biological Availability; 1-Deoxynojirimycin
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — miglustat

INTERVENTIONS:
Drug: Butyldeoxynojirimycin

SUMMARY:
To determine the following about the use of SC-48334 in patients with AIDS and advanced AIDS related complex (ARC):

1. The largest maximum tolerated dose (MTD); 2. Effectiveness against HIV; 3. Pharmacokinetics - how fast SC-48334 reaches the bloodstream, what concentration is reached, and how long it remains in the patient's blood.

SC-48334 is a chemical that prevents the biochemical actions of certain enzymes in the body, and recent studies have shown that it may also prevent the activity of HIV. The study will attempt to show whether SC-48334 can safely and effectively break the cycle of HIV infection in AIDS and advanced ARC by progressively eliminating HIV.

DETAILED DESCRIPTION:
SC-48334 is a chemical that prevents the biochemical actions of certain enzymes in the body, and recent studies have shown that it may also prevent the activity of HIV. The study will attempt to show whether SC-48334 can safely and effectively break the cycle of HIV infection in AIDS and advanced ARC by progressively eliminating HIV.

Six patients are enrolled sequentially into each of eight different dose levels and the drug is administered by mouth at least 60 minutes before meals according to the following schedule: Day 1: One-quarter of total assigned daily dose. Patients receive the dosage in the hospital as either an inpatient or outpatient and are observed for 12 hours, during which time they are evaluated and blood is drawn for pharmacokinetic studies. Patients return at 24 and 48 hours for a limited physical examination and additional pharmacokinetic studies. Days 4 - 31: Total assigned daily dose, one-quarter 4 times a day. Patients are observed for at least 5 days in the hospital following the start of this part of the program, during which time clinical, laboratory, and pharmacokinetic information is obtained in order to establish baseline values. After the 6th day, patients are evaluated with a complete physical exam, urinalysis, and laboratory studies once a week and a limited physical exam and brief laboratory studies 3 times a week. At each of the eight dose levels, the second and third patients receive their first dose only after the first patient has been followed for 72 hours after receiving the first dose. Patients 4, 5, and 6 begin treatment only after patients 2 and 3 have completed 14 days of the four-part total dose. Patients are treated on an outpatient basis, with 5 to 6 days spent in the hospital for evaluation.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine.
* Nystatin.
* Clotrimazole.
* Topical acyclovir.

Concurrent Treatment:

Allowed:

* Blood transfusions for = or > grade 3 hemoglobin toxicity.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions will be excluded:

* Clinical significant diarrhea (> 3 stools per day for > 7 days without definable cause).
* Active opportunistic infection, requiring ongoing therapy, at time of enrollment.
* Any malignancy besides Kaposi's sarcoma, basal cell carcinoma, or squamous cell carcinoma unless the squamous cell carcinoma requires ongoing therapy.
* Neurologic disease including dementia, peripheral neuropathy, myelopathy (CDC category IVb).

Concurrent Medication:

Excluded:

* Antimetabolites.
* Alkylating agents.
* Drugs with known hepatic or bone marrow toxicity.

Patients with significant organ dysfunction will be excluded.

Prior Medication:

Excluded:

* Antimetabolites.
* Alkylating agents.
* Excluded within 30 days of study entry:
* Any investigational medication.
* Drugs with anti-HIV activity.
* Excluded within 90 days of study entry:
* Ribavirin treatment.
* Excluded within 6 months of study entry:
* Cancer chemotherapy.

Prior Treatment:

Excluded within 6 months of study entry:

* Radiation therapy.

Patients must demonstrate the following clinical and laboratory findings:

* AIDS or advanced AIDS related complex (ARC), according to Centers for Disease Control (CDC) category IV, excluding neurologic disease in IVb.
* Ability to understand the terms of study participation.

Current use of illicit drugs or abuse of alcohol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48

CONTACTS AND LOCATIONS:
Overall Officials: MS Hirsch, Study Chair
Locations (6):
- United States (6):
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Stanford Univ School of Medicine, Stanford, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Julio Arroyo, West Columbia, South Carolina

REFERENCES:
- [Background] Tierney M, Pottage J, Kessler H, Fischl M, Richman D, Merigan T, Powderly W, Smith S, Karim A, Sherman J, et al. The tolerability and pharmacokinetics of N-butyl-deoxynojirimycin in patients with advanced HIV disease (ACTG 100). The AIDS Clinical Trials Group (ACTG) of the National Institute of Allergy and Infectious Diseases. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Dec 15;10(5):549-53. PMID 8548334